CLINICAL TRIAL: NCT03553368
Title: Chest Imaging of Lung Nodule(s) Under High-frequency Non-invasive Ventilation (HF-NIV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Beigelman-Aubry Catherine, PD-MER, Head of the Chest Imaging Unit, University of Lausanne Hospitals
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: HF-NIV-MR-PET
Record Dates: First submitted 2018-05-15; First posted 2018-06-12 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Neoplasms
Keywords: lung nodules
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Step 1: Healthy volunteers (Experimental): Experimental intervention:
  MRI data will be acquired with the use of HF-NIV (HF-NIV-MR).
  Control intervention:
  MRI data will be acquired without the use of HF-NIV, as a reference (MR).
  Interventions: Diagnostic Test: HF-NIV-MR; Diagnostic Test: MR
- Step 2: Patients (arm A) (Experimental): Experimental intervention:
  MRI data will be acquired with the use of HF-NIV (HF-NIV-MR).
  Control intervention:
  MRI data will also be acquired without the use of HF-NIV, as a reference (MR). The clinically prescribed CT will be the gold standard.
  Interventions: Diagnostic Test: HF-NIV-MR; Diagnostic Test: MR
- Step 2: Patients (arm B) (Experimental): Experimental intervention:
  PET/CT data will be acquired with the use of HF-NIV (HF-NIV-PET). MRI data will be acquired with the use of HF-NIV (HF-NIV-MR). PET/CT data will be acquired in inspiratory breath hold without the use of HF-NIV (PET/CT breath hold).
  Control intervention:
  Data from the clinically indicated PET/CT acquisition will be used as reference.
  MRI data will also be acquired without the use of HF-NIV, as a reference (MR). Histological data will be used when available.
  Interventions: Diagnostic Test: HF-NIV-MR; Diagnostic Test: HF-NIV-PET; Diagnostic Test: MR; Diagnostic Test: PET/CT breath hold
- Step 1 bis: Healthy volunteers (Experimental): Experimental intervention:
  MRI data will be acquired with the use of CPAP (CPAP-MR).
  Control intervention:
  MRI data will be acquired without the use of CPAP, as a reference (MR).
  Interventions: Diagnostic Test: MR; Diagnostic Test: CPAP-MR

INTERVENTIONS:
Diagnostic Test: HF-NIV-MR — MRI data will be acquired with the use of HF-NIV.
  Arms: Step 1: Healthy volunteers; Step 2: Patients (arm A); Step 2: Patients (arm B)
Diagnostic Test: HF-NIV-PET — PET data will be acquired with the use of HF-NIV.
  Arms: Step 2: Patients (arm B)
Diagnostic Test: MR — MRI data will be acquired without the use of any device as a reference.
Diagnostic Test: PET/CT breath hold — PET/CT data will be acquired in inspiratory breath hold without the use of HF-NIV.
  Arms: Step 2: Patients (arm B)
Diagnostic Test: CPAP-MR — MRI data will be acquired with the use of CPAP.
  Arms: Step 1 bis: Healthy volunteers

SUMMARY:
Imaging of chest disorders is mainly achieved by using computed tomography. This is especially the case for detection, morphologic assessment and followup of pulmonary nodules. A positron emission tomography (PET) /CT may be additionally required for lung nodule management in some conditions including a size greater than 8 mm with morphologic or growing characteristics suspicious of malignancy. Magnetic Resonance Imaging (MRI) represents however an interesting alternative diagnostic radiation-free method, in particular owing to the recent development of sequences dedicated to lung parenchyma analysis. A major limitation remains the control of respiratory artefacts.

High Frequency non-invasive ventilation, HF-NIV, has the potential to allow chest stabilization and is currently used in the department of radio-oncology at the Lausanne University Hospital. It has been recently applied to perform MRI and PET examinations at end inspiration during an "apnea " generated by the system. Continuous periods of respiratory stabilization of several minutes at end-inspiration are thus obtained, allowing prolonged MR and PET acquisitions with improvement of image quality as observed in our preliminary studies (Beigelman-Aubry et al., Prior et al.). Interestingly, the lung volume explored by using this ventilation technique is similar to that of CT studies, conversely to respiratory gated MR sequences which are currently performed at end-expiration, this potentially generating underevaluation of lung disorders especially at lung bases.

The present project aims to determine the impact of HF-NIV in the management of patients with pulmonary nodule(s). After a first step of optimization of acquisition parameters of HF-NIV-MR in healthy volunteers, the performances of MRI and PET/CT (when required) under this ventilation technique will be compared to the current method(s) of reference in cases of pulmonary nodule(s) (CT scan and PET when required) and histological data when available. All MRI and PET/CT (when required) acquisitions will be performed without the ventilation technique, as used in current practice, and with it.

The project was completed with an amendment to investigate MRI under continuous positive airway pressure (CPAP). The MR-CPAP combination will be evaluated with optimized parameters in healthy volunteers and compared to free-breathing acquisitions without any device.

ELIGIBILITY:
Inclusion Criteria:

* Validated Informed Consent as documented by signature (Appendix Informed Consent Form)
* Depending on study arm:
* Good health (step 1 and 1 bis only) or
* Patients with at least 1 non calcified pulmonary nodule of at least 4 mm, whatever its texture (solid, sub-solid) and nature (benign, indeterminate or malignant), just discovered or in a follow-up context (step 2 only)
* Age ≥ 18 years

Exclusion Criteria:

* Previous or current disorder that might interfere with performance or safety of study procedures
* Age <18 years
* Any contraindication to MRI (pace makers, neuro-stimulators, some implantable devices, some metallic implants, claustrophobia)
* Any contraindication to a positive airway pressure therapy (claustrophobia, fracture of the skull, right heart failure), (step 1 bis)
* Children, adolescents and adults with incapacities
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Pregnant or breastfeeding women
* Chronic obstructive pulmonary disease (COPD) or asthma with severe obstruction

  * Severe obstructive patients (FEV1<50% of predicted value)
  * Hypoxemia (SaO2<94% AA)
  * History or physical signs of right heart failure
* History or physical signs of right or left cardiac failure
* History or physical signs of pulmonary hypertension
* History or physical signs of active coronary artery disease
* Pulmonary graft
* Immunocompromized patients
* Enrollment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Image quality, step 1: Healthy volunteers, sharpness of vessels | day 1
  Sharpness of interfaces of vessels will be scored on a discrete scale as 1=blurred; 2=intermediate; 3=sharp. This will determine the adequate choice of MR sequences and parameters.
Sensitivity for nodule detection, step 2: Patients (arm A) | day 1
  Determine whether HF-NIV-MR allows a better detection (higher sensitivity) of the presence of pulmonary nodules compared with conventional MR. CT will be used as gold standard.
Sensitivity for nodule characterization, step 2: Patients (arm B) | day 1
  Determine whether sensitivity of the apparent diffusion coefficient (ADC) value obtained with HF-NIV-MR (diffusion sequence) to characterize nodules is higher than the sensitivity obtained with conventional MRI. Histological data will be used as gold standard when available.
Assessment of CPAP-MR, step 1 bis: Healthy volunteers | day 1
  Determine whether CPAP-MR has an additional value compared with MR. Image quality of the CPAP-MR acquisition will be evaluated similarly to the methodology of step 1 and compared to the gold standard MR acquisition (free-breathing without any device).

SECONDARY OUTCOMES:
Image quality, step 1: Healthy volunteers, sharpness of bronchi | day 1
  Sharpness of interfaces of bronchi will be scored on a discrete scale as 1=blurred; 2=intermediate; 3=sharp.
Image quality, step 1: Healthy volunteers, sharpness of fissures | day 1
  Sharpness of interfaces of fissures will be scored on a discrete scale as 1=blurred; 2=intermediate; 3=sharp.
Image quality, step 1: Healthy volunteers, visibility of vessels | day 1
  Modified criteria of Ohno (Ohno et al.) will be used and vessels will be scored as follows 0=non visible; 1=depicted at a lobar level; 2=depicted at a segmental level; 3=depicted at a sub-segmental level; 4=depicted at a sub-sub segmental level; 5=depicted beyond the sub-subsegmental level.
Image quality, step 1: Healthy volunteers, visibility of bronchi | day 1
  Modified criteria of Ohno (Ohno et al.) will be used and bronchi will be scored as follows 0=non visible; 1=depicted at a lobar level; 2=depicted at a segmental level; 3=depicted at a sub-segmental level; 4=depicted at a sub-sub segmental level; 5=depicted beyond the sub-subsegmental level.
Image quality, step 1: Healthy volunteers, visibility of fissures | day 1
  Fissures will be scored as follows 0=non visible; 1=visible.
Nodule dimensions | day 1
  The variable of interest will be the volumetry of each nodule detected which will be evaluated by using dedicated software. This will be compared with volumetric assessment by using CT performed less than 1 month before the MR examination, at best the same day.
  Two-Dimensional measurements (long axis, mean of the long and short diameter) will also be used, in accordance with usual recommendations [MacMahon et al.].
MR-PET fusion | day 1
  Fusion of MR acquisitions and PET under HF-NIV should be obtained with a good accuracy. The correspondence will be evaluated with a fiducial anatomical structures technique, as if acquisitions were done on a PET-MR scanner.
Correlation of diffusion MRI with metabolic activity | day 1
  The correlation between ADC (diffusion coefficient) and metabolic activity in HF-NIV-PET/CT, will be compared to the one obtained without HF-NIV.
PET/CT stabilization assessment | day 1
  The PET/CT image stabilization methods will compared and the best one will be determined (electronic respiratory-gating during the normal free-breathing PET/CT, a single short PET/CT apnea (<30 seconds) and the HF-NIV-PET/CT acquisition.
Correlation with ex-vivo nodule volume | day 1
  When applicable, the volume of lesions measured on imaging studies will be compared to the volume measured ex-vivo following surgical resection.
Tolerance CPAP-MR, step 1 bis: Healthy volunteers | day 1
  Subject subjective tolerance to CPAP-MR will be scored on a 5 points discrete scale as follows: 0=no additional discomfort, 1=minor discomfort, 2=moderate discomfort, 3=high discomfort, 4=extreme discomfort (same methodology as for steps 1 and 2).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Beigelman-Aubry, MD, Principal Investigator — University Hospital Lausanne (CHUV), Radiology
Locations (1):
- University Hospitals, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beigelman-Aubry C, Peguret N, Stuber M, Delacoste J, Belmondo B, Lovis A, Simons J, Long O, Grant K, Berchier G, Rohner C, Bonanno G, Coppo S, Schwitter J, Ozsahin M, Qanadli S, Meuli R, Bourhis J. Chest-MRI under pulsatile flow ventilation: A new promising technique. PLoS One. 2017 Jun 12;12(6):e0178807. doi: 10.1371/journal.pone.0178807. eCollection 2017. PMID 28604833
- [Background] Prior JO, Peguret N, Pomoni A, Pappon M, Zeverino M, Belmondo B, Lovis A, Ozsahin M, Vienne M, Bourhis J. Reduction of Respiratory Motion During PET/CT by Pulsatile-Flow Ventilation: A First Clinical Evaluation. J Nucl Med. 2016 Mar;57(3):416-9. doi: 10.2967/jnumed.115.163386. Epub 2015 Dec 3. PMID 26635339
- [Background] MacMahon H, Naidich DP, Goo JM, Lee KS, Leung ANC, Mayo JR, Mehta AC, Ohno Y, Powell CA, Prokop M, Rubin GD, Schaefer-Prokop CM, Travis WD, Van Schil PE, Bankier AA. Guidelines for Management of Incidental Pulmonary Nodules Detected on CT Images: From the Fleischner Society 2017. Radiology. 2017 Jul;284(1):228-243. doi: 10.1148/radiol.2017161659. Epub 2017 Feb 23. PMID 28240562
- [Background] Ohno Y, Koyama H, Yoshikawa T, Seki S, Takenaka D, Yui M, Lu A, Miyazaki M, Sugimura K. Pulmonary high-resolution ultrashort TE MR imaging: Comparison with thin-section standard- and low-dose computed tomography for the assessment of pulmonary parenchyma diseases. J Magn Reson Imaging. 2016 Feb;43(2):512-32. doi: 10.1002/jmri.25008. Epub 2015 Jul 30. PMID 26223818
- [Result] Darcot E, Delacoste J, Dunet V, Dournes G, Rotzinger D, Bernasconi M, Vremaroiu P, Simons J, Long O, Rohner C, Ledoux JB, Stuber M, Lovis A, Beigelman-Aubry C. Lung MRI assessment with high-frequency noninvasive ventilation at 3 T. Magn Reson Imaging. 2020 Dec;74:64-73. doi: 10.1016/j.mri.2020.09.006. Epub 2020 Sep 6. PMID 32898653